CLINICAL TRIAL: NCT06512636
Title: A Decade-Long Dance With Diplopia: Unraveling the Enigma of Recurrent 6th Nerve Palsy
Status: Completed | Type: Observational
Sponsor: College of Medical Sciences, Bharatpur (Other)
Responsible Party: Principal Investigator, Kamal Raj Baral, Doctor, College of Medical Sciences, Bharatpur
Other Study IDs: 0000
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Neurologic Manifestations
MeSH Terms: conditions — Neurologic Manifestations

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Abstract:

Introduction and Importance:

Recurrent diplopia poses a diagnostic challenge, necessitating a thorough evaluation to elucidate its underlying etiology and guide its management. We present the case of a 39-year-old farmer with recurrent 6th nerve palsy for over a decade, highlighting the complexity and persistence of this condition.

Case Presentation:

A 39-year-old farmer presented with recurrent diplopia attributed to 6th nerve palsy, with eight episodes over 14 years. Despite systemic steroid treatment, the symptoms recurred every 12-18 months. Clinical examination revealed right eye abduction impairment;-, no other abnormalities were detected. Magnetic resonance imaging (MRI) indicated rhinosinusitis, and the results of the autoimmune antibody test were negative.

Clinical Discussion:

This case challenges conventional diagnostic approaches, underscoring the need for a comprehensive evaluation and tailored management strategies. Despite extensive investigations, the etiology remains elusive, emphasizing the complexity of recurrent diplopia.

Conclusion:

Continued monitoring and further investigation are warranted to unravel the enigma of recurrent diplopia in this unique case, highlighting the importance of individualized approaches to guide optimal management.

DETAILED DESCRIPTION:
A Decade-Long Dance with Diplopia: Unraveling the Enigma of Recurrent 6th Nerve Palsy

ABSTRACT

Introduction and Importance:

Recurrent diplopia poses a diagnostic challenge, necessitating a thorough evaluation to elucidate its underlying etiology and guide its management. We present the case of a 39-year-old farmer with recurrent 6th nerve palsy for over a decade, highlighting the complexity and persistence of this condition.

Case Presentation:

A 39-year-old farmer presented with recurrent diplopia attributed to 6th nerve palsy, with eight episodes over 14 years. Despite systemic steroid treatment, the symptoms recurred every 12-18 months. Clinical examination revealed right eye abduction impairment;-, no other abnormalities were detected. Magnetic resonance imaging (MRI) indicated rhinosinusitis, and the results of the autoimmune antibody test were negative.

Clinical Discussion:

This case challenges conventional diagnostic approaches, underscoring the need for a comprehensive evaluation and tailored management strategies. Despite extensive investigations, the etiology remains elusive, emphasizing the complexity of recurrent diplopia.

Conclusion:

Continued monitoring and further investigation are warranted to unravel the enigma of recurrent diplopia in this unique case, highlighting the importance of individualized approaches to guide optimal management.

Keywords: Recurrent diplopia, 6th nerve palsy, autoimmune disease, systemic steroid, neuro-ophthalmology.

Highlights

* Recurrent diplopia is a diagnostic puzzle, especially in terms of etiology
* Despite treatment, the patient experienced recurrent diplopia attributed to 6th nerve palsy for 14 years, highlighting the chronic nature of the condition.
* Extensive evaluation failed to identify the underlying cause, which illustrates the diagnostic complexity of recurrent diplopia.
* Systemic steroid treatment provided temporary relief, but the recurrence persisted, necessitating long-term management.
* This case emphasizes the need for tailored approaches and ongoing monitoring to effectively address the challenges in managing recurrent diplopia.

INTRODUCTION Recurrent diplopia presents a diagnostic problem, especially when associated with 6th nerve palsy. The etiology of recurrent diplopia in older individuals has yet to be well described in the literature.1 We present a case of a 39-year-old male farmer with eight episodes of diplopia over 14 years, each responding to systemic steroid therapy but recurring every 12-18 months. Despite the patient's clinical response, the underlying etiology remains elusive, emphasizing the complexity of this rare condition. This case prompts a thorough exploration of the potential inflammatory or autoimmune origins of recurrent 6th nerve palsy, addressing the disorder's symptomatic relief and recurrent nature.1,2 This report contributes to the limited literature on such cases, shedding light on the challenges and considerations in managing this recurrent neuro-ophthalmological condition.

CASE REPORT

In this case, a 39-year-old male, a married farmer, was presented to the Neuromedicine OPD for a follow-up examination of recurrent diplopia attributed to 6th nerve palsy. The patient reported no recent instances of double vision or associated complaints during the follow-up visit. Notably, the last episode of diplopia occurred 13 months prior, and the patient had experienced eight such episodes over 14 years since 2008.

During the previous episode, the patient sought medical attention with the chief complaint of acute-onset double vision persisting for 10 days. No significant concurrent medical or surgical issues were reported, aside from a recurrent history of diplopia, and treatment during previous occurrences involving systemic steroid administration, resulting in the complete resolution of symptoms. Recurrence typically manifest within 12-18 months of treatment.

Clinical examination revealed that the patient could not abduct the right eye, whereas the remaining ocular and systemic examinations yielded normal results. Notably, there were no signs of myasthenia gravis, ptosis, and pain on the movement of the eyeballs, decreased visual acuity, trauma, red eyes, headache, focal neurological deficits, or meningeal or cerebellar abnormalities. Brain MRI revealed no abnormalities, except for the presence of rhinosinusitis.

A comprehensive antibody panel, including anti-acetylcholinesterase receptor antibodies and anti-MUSK antibody tests, was used to investigate the possibility of an autoimmune etiology. All results from these tests were negative, further complicating the determination of the underlying cause of recurrent diplopia. Continued monitoring and further investigations may be necessary to elucidate the nature of this unique case and to guide appropriate management.

DISCUSSION

The case of a 39-year-old male farmer with recurrent diplopia attributed to 6th nerve palsy highlights the diagnostic challenges and complexities of managing this rare condition. Despite the patient's clinical response to systemic steroid therapy, the underlying etiology remains elusive, emphasizing the need for thorough exploration of the potential inflammatory or autoimmune origins of recurrent 6th nerve palsy.

The literature suggests that benign recurrent 6th nerve palsy in children is rare, and recurrences are rarer.3, 4 This condition typically occurs following viral illnesses, infections, and immunization involving attenuated live vaccinations. In adults, the evaluation and management of recent-onset diplopia in adults with a history of long-standing strabismus can be perplexing and challenging.5 The causes of isolated recurrent ipsilateral sixth nerve palsies in older adults have not been well described in the literature, and the etiology of recurrent isolated sixth nerve palsies in older adults has not been well described.1 The clinical presentation of isolated recurrent diplopia from a sixth nerve palsy should prompt a neurologist or ophthalmologist to order a brain MRI with and without gadolinium as part of the initial workup to rule out a non-microvascular cause, such as a compressive lesion.1 The exact pathophysiologic mechanism of the relapsing and remitting course of the sixth nerve palsy has yet to be fully understood. This may be related to a structural lesion or an inflammatory process.1 The etiological diagnosis of diplopia is a clinical challenge.4 Binocular diplopia is referred to in the literature as the most common type, and there are several etiological mechanisms of binocular diplopia, including orbital disorders, extra-ocular muscle disorders, neuromuscular junction dysfunction, and primary or secondary visual cortex diseases.4 In conclusion, the case of a 39-year-old male farmer with recurrent diplopia attributed to 6th nerve palsy highlights the diagnostic challenges and complexities of managing this rare condition. The literature suggests that benign recurrent 6th nerve palsy in children is rare, and recurrences are rarer. By contributing to the existing literature on this rare condition, we aimed to enhance awareness among clinicians and foster a multidisciplinary approach to patient care, ultimately improving outcomes in individuals with similar presentations.

Consent:

Written informed consent was obtained from the patient for the publication of this case report. A copy of the written consent form is available for review by the editor-in-chief of the journal upon request.

Ethical Approval:

Ethical approval is not required for case report.

Source of Funding:

There is no source of Funding.

Research Registration:

Research registration is not required as this is only a case report.

Author contribution:

P.P.: Conceptualization, project administration, supervision, writing -review, and editing. K.R.B.: Conceptualization, project administration, supervision, writing-review, and editing. R.K.C: Formal analysis, writing -original draft, writing-review, and editing. N.R.: Writing- original draft, writing-review and editing. S.M.: Resources, supervision, writing-original draft, writing-review and editing. B.A.: Resources, writing-original draft, writing-review, and editing. K.S.: Resources, writing-original draft, writing-review, and editing.

Conflict of Interest:

The authors declare that they have no conflicts of interest. The work has been reported as being in line with SCARE criteria.

Guarantor:

Prabesh Panta.

Data availability statement:

The datasets are available from the corresponding author on reasonable request.

REFERENCES:

1. Chan JW, Albretson J. Causes of isolated recurrent ipsilateral sixth nerve palsies in older adults: a case series and review of the literature. Clin Ophthalmol Auckl NZ. 2015;9:373. Available from: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4348047/
2. Patel SV, Mutyala S, Leske DA, Hodge DO, Holmes JM. Incidence, associations, and evaluation of sixth nerve palsy using a population-based method. Ophthalmology. 2004 Feb ;111(2):369-75. Available from: https://linkinghub.elsevier.com/retrieve/pii/S0161642003011849
3. Gonçalves R, Coelho P, Menezes C, Ribeiro I. Benign Recurrent Sixth Nerve Palsy in a Child. Case Rep Ophthalmol Med. 2017:8276256. Available from: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5763058/
4. Kushner BJ. Recently Acquired Diplopia in Adults With Long-standing Strabismus. Arch Ophthalmol. 2001 Dec 1;119(12):1795-801. Available from: https://doi.org/10.1001/archopht.119.12.1795
5. Alves M, Miranda A, Narciso MR, Mieiro L, Fonseca T. Diplopia: A Diagnostic Challenge with Common and Rare Etiologies. Am J Case Rep. 2015 Apr 13;16:220-3. Available from: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4410729/

ELIGIBILITY:
Inclusion Criteria:

* This is only a case report of 39-years-old male.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a case report of a 39 year old male.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
A Decade-Long Dance with Diplopia: Unraveling the Enigma of Recurrent 6th Nerve Palsy | 6 months
  As this is only a case report. No primary outcome was present.

CONTACTS AND LOCATIONS:
Overall Officials: Prabesh Panta, Principal Investigator — College of Medical Sciences, Bharatpur
Locations (1):
- Kamal Raj Baral, Bharatpur, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: Undecided
This is a case report only and we are trying to obtain the Rrsearch registration ID. If the Clinicaltrials.gov need more information about this case report then feel free to contact at kamalrajbaral74@gmail.com